CLINICAL TRIAL: NCT01122160
Title: Gastric pH as a Possible Determinant of Anthocyanin Absorption
Brief Title: Gastric pH and Anthocyanin Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 2010-069
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-07

CONDITIONS: Anthocyanin Metabolism
Keywords: anthocyanin; omeprazole; Prilosec; gastric pH; proton pump inhibitor; PPI; nutrition
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Placebo with berries (blackberries + strawberries)
  Interventions: Drug: placebo
- omeprazole (Experimental): Prilosec (omeprazole) 20.6 mg tablet with berries (blackberries + strawberries)
  Interventions: Drug: omeprazole

INTERVENTIONS:
Drug: omeprazole — omeprazole 20.6 mg tablet with berries (blackberries + strawberries)
  Arms: omeprazole
Drug: placebo — Placebo with berries (blackberries + strawberries)
  Arms: placebo

SUMMARY:
Anthocyanins are phytonutrients that provide blue, purple and red colors to fruits and vegetables. The purpose of the study is to determine whether absorption of anthocyanins occurs in the acid pH of the stomach and to determine whether altering stomach pH by use of an over-the-counter medicine, Prilosec TM, alters absorption of anthocyanins from strawberries and blackberries.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 kg/m2 to 30 kg/m2
* Age 22 to 59 years

Exclusion Criteria:

* Plans to have MRI analysis or other contact with MRI equipment during the study
* Has implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump
* Suspected strictures, fistulas or physiological GI obstruction
* Allergy to omeprazole
* Current use of clopidogrel (Plavix) or use within the past 3 months
* Use of warfarin, prescription antifungals/anti-yeast drugs, diazepam, and digoxin
* Chronic daily use of nonsteroidal anti-inflammatory drugs (ibuprofen, naproxen, etc.)
* History of bariatric or other gastric surgery
* Frequent use of antacids
* Use of proton pump inhibitors in past 3 months
* History of acid reflux
* History of gastrointestinal disorders or gastrointestinal surgery
* History of bezoars (packed collection of partially digested or undigested material that is unable to exit the stomach)
* Crohn's disease, diverticulitis or inflammatory bowel disease
* Inability to swallow large pills
* Dysphagia (Trouble or pain with swallowing food or pills)
* Allergy to strawberries or blackberries
* Pregnant women
* Lactating women
* Pregnancy in last 12 months
* History of kidney disease
* History of liver disease
* History of metabolic disorder
* History of some cancers
* Tobacco use in past 6 months
* Use of oral or IV antibiotics in past month
* Use of herbal supplement in past month

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Clevidence, Ph. D., Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA's Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Discrepancy between actual enrollment and number of participants in participant flow module is due to enrolled participants no longer meeting exclusion criteria (i.e., inability to swallow capsule).
Groups:
- Placebo First, Then Omeprazole: Placebo with berries (blackberries + strawberries), followed by Omeprazole with berries (blackberries + strawberries)
- Omeprazole First, Then Placebo: Prilosec (omeprazole) 20.6 mg tablet with berries (blackberries + strawberries), followed by placebo with berries (blackberries + strawberries)
Period: First Intervention (7 Days)
Arm/Group | Placebo First, Then Omeprazole | Omeprazole First, Then Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (7-14 Days)
Arm/Group | Placebo First, Then Omeprazole | Omeprazole First, Then Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Placebo First, Then Omeprazole | Omeprazole First, Then Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants received both interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Gastric pH
Time Frame: 1 hour prior to gastric emptying on Day 7 of the given intervention
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 11 | 11
pH | 0.96 (0.37) | 2.31 (0.63)

ADVERSE EVENTS:
Arm/Group | Experimental | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes